CLINICAL TRIAL: NCT04064372
Title: Mindful Response to Adversity: A Brief Stress Resilience Training for Improving Mental Health in Students
Brief Title: Mindful Response to Adversity: A Brief Stress Resilience Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 182R07SM
Record Dates: First submitted 2019-01-01; First posted 2019-08-21 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Loneliness; Depression
Keywords: Mindfulness; Resilience; Equanimity; Inflammation; Wise Intervention
MeSH Terms: conditions — Depression; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will remain masked to which program the participant will use. However the experimenter will engage with participants while in their training groups and thus will not be masked to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Response to Adversity (Experimental): The treatment condition will be trained in techniques designed to teach a "mindful approach to adversity". These techniques will include: normalizing, attention, equanimity, non-judgment, de-centering, accepting of experiences, and impermanence. Participants will be instructed on the mindset, asked to write about an instance of non-judgment and share with a partner, and then guided through a short training designed to practice each skill.
  Interventions: Behavioral: Mindful response to adversity brief training
- Strength-based approach to adversity (Active Comparator): The control condition will be trained in techniques designed to teach a typical narrative self-analysis / strengths-based approach to adversity. These techniques will include: choosing the best approach, minimizing stress, and identifying and enhancing personal strengths. Participants will be instructed on the mindset, asked to write about an instance of personal strength and share with a partner, and then guided through a short training designed to practice each skill.
  Interventions: Behavioral: Strengths-based response to adversity brief training

INTERVENTIONS:
Behavioral: Mindful response to adversity brief training — Participants will attend a group training session, led by a professional instructor, about responding to adversity with an approach of mindfulness, equanimity, and non-judgment, which will include a description of the skills, a writing and sharing activity focused on the proposed approach, and a practice session. Following the training, participants will be instructed to practice the skills that they just learned during a group version of a standard stress-induction task called the Trier Social Stress Task (the TSST-G).
  Arms: Mindful Response to Adversity
Behavioral: Strengths-based response to adversity brief training — Participants will attend a group training session, led by a professional instructor, about responding to adversity with an approach of strengths-based, narrative self-analysis, which will include a description of the skills, a writing and sharing activity focused on the proposed approach, and a practice session. Following the training, participants will be instructed to practice the skills that they just learned during a group version of a standard stress-induction task called the Trier Social Stress Task (the TSST-G).
  Arms: Strength-based approach to adversity

SUMMARY:
The investigators will conduct an intervention study with the aim of improving stress resilience and mental health outcomes in at-risk freshman students. Participants will attend a group training session, led by a professional instructor, about responding to adversity, which will include a description of the skills, a writing and sharing activity focused on the proposed approach, and a practice session. Following the training, participants will be instructed to practice the skills that the participants just learned during a group version of a standard stress-induction task called the Trier Social Stress Task (the TSST-G).

DETAILED DESCRIPTION:
The investigators will conduct an intervention study with the aim of improving stress resilience and mental health outcomes in at-risk freshman students. The investigators will also work closely with institutional officials to assess whether the intervention can improve student well-being. Specifically, the project aims to teach freshman students (who are at high risk for depression) skills in how to foster a mindful response to adversity at the beginning of the school term, along with periodic support reminders (via text message) during high stress/vulnerability periods over the course of the semester. The investigators will adopt a randomized controlled trial approach to rigorously evaluate whether this intervention can be adopted as a standard onboarding program for all incoming freshman students during the first weeks of orientation on the CMU campus. Participants will come for the study session and provide a dried blood spot sample and complete a battery of self-report questionnaires.

Participants will attend a group training session, led by a professional instructor, about responding to adversity, which will include a description of the skills, a writing and sharing activity focused on the proposed approach, and a practice session. Following the training, participants will be instructed to practice the skills that the participants just learned during a group version of a standard stress-induction task called the Trier Social Stress Task (the TSST-G). Salivary cortisol measures will be collected throughout the TSST-G.

The treatment condition will be trained in techniques designed to teach a "mindful approach to adversity". These techniques will include: normalizing, attention, equanimity, non-judgment, de-centering, accepting of experiences, and impermanence. Participants will be instructed on the mindset, asked to write about an instance of non-judgment and share with a partner, and then guided through a short training designed to practice each skill.

The control condition will be trained in techniques designed to teach a typical narrative self-analysis / strengths-based approach to adversity. These techniques will include: choosing the best approach, minimizing stress, and identifying and enhancing personal strengths. Participants will be instructed on the mindset, asked to write about an instance of personal strength and share with a partner, and then guided through a short training designed to practice each skill.

Daily diary measures will be collected for 7 days following the study session and 1 week before the follow-up session. Microhit boosters will be sent to participants at self-identified high stress periods, which remind participants of the training session skills.

Participants will come for the follow-up session and provide a dried blood spot sample and complete a battery of self-report questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Full-time first-year student at Carnegie Mellon University.
* Adult (age 18+)
* Must own a data-enabled smartphone
* Scores indicating moderate to high levels of depressive symptomatology (composite score > or equal to 2 on the short-form (6-item) Beck Depression Inventory).

Exclusion Criteria:

* Potential participants who score a 0 or a 1 on the 6-item BDI section will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Daily Depression | Change in daily depression assessed daily for seven days during week 2 and week 16 of the study.
  In a daily diary, participants are asked at the end of the day to identify the extent to which they endorse symptoms measuring depressive symptomatology (i.e. "feeling hopeless about the future", "feeling blue") for that day.
  Analyses will use multilevel modeling to test for a time by condition interaction showing lower daily depressive symptomatology at post-treatment in the equanimity compared to the strength based group.
Depression I | Change in depression over 4-month period.
  Evaluated using the validated 21-item Beck Depression Inventory (BDI), which is designed to measure characteristic attitudes and symptoms of depression. The score for each item ranges between 0-3, where 0 denotes less depression (e.g. "I do not feel sad") and 3 denotes more depression (e.g. "I am so dan and unhappy that I can't stand it"). Total score will be between 0-63, where 0 indicates no depression and 63 indicates extreme depression. The score is a total of 21 questions and the following is a typical subscale range distribution:
  1-10: These ups and downs are considered normal 11-16: Mild mood disturbance 17-20: Borderline clinical depression 21-30: Moderate depression 31-40: Severe depression over 40: Extreme depression Analyses will use multilevel modeling to test for a time by condition interaction showing lower depressive symptomatology at post-treatment in the equanimity compared to the strength based treatment group.
Depression II | Change in depression over 4-month period.
  Evaluated using the validated 20-item Center for Epidemiologic Studies Depression scale (CES-D), which is designed to measure characteristic attitudes and symptoms of depression. There are 20 questions and the score for each item ranges between 0-3. For most questions, a lower score indicates lack of depression and a higher score indicates high depression (e.g. in response to the statement "I felt fearful" a 0 indicates rarely and 3 indicates most or all of the time). Questions 4, 8, 12, and 16 are reverse scored. The score is the sum of the 20 questions. Possible range is 0-60. A score of 16 points or more is considered depressed.
  Analyses will use multilevel modeling to test for a time by condition interaction showing lower depressive symptomatology at post-treatment in the equanimity compared to the strength based treatment group.
Daily Social Connection | Change in daily social connection assessed daily for seven days during week 2 and week 16 of the study.
  Following Hawkley et al. (2007) and our previous studies, end-of-day daily diary questions will assess the amount of time spent interacting with others and the extent to which social interactions throughout the day were perceived as positive. Example items: "How much time did you spend today with others, talking or listening to them?" (0 = little or none of the day to 4 = most or all of the day) and "How many positive interactions did you have today (e.g., supportive, enjoyable, rewarding, affirming)?" (0 = one, 1 = several, 2 = many).
  Analyses will use multilevel modeling to test for a time by condition interaction showing increased daily social connection at post-treatment in the equanimity compared to the strength based group.
Daily Belonging | Change in loneliness over 4-month period.
  End-of-day daily diary questions will measure feelings of belonging and closeness at school. Example items: "I felt like I belong in school" and "I felt like no one really knew me well at school (reverse-scored)" (0= Not at all, 4= Extremely).
  Analyses will use multilevel modeling to test for a time by condition interaction showing increased daily social belonging at post-treatment in the equanimity compared to the strength based group.
Loneliness | Change in loneliness over 4-month period.
  Evaluated using the University of California, Los Angeles (UCLA) Loneliness Scale. The University of California, Los Angeles (UCLA) Loneliness scale is designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as either A ("I always feels this way"), O ("I often feel this way"), S ("I sometimes feel this way"), R ("I rarely feel this way"), N ("I never feel this way"). Scores are summed from each item and higher scores indicate greater degrees of loneliness. Scores of 15-20 indicate average level of loneliness; 21-30 indicate frequent loneliness; 31-40 indicate severe loneliness.
  Analyses will use multilevel modeling to test for a time by condition interaction showing decreased loneliness at post-treatment in the equanimity compared to the strength based group.

SECONDARY OUTCOMES:
Academic performance | Change in GPA between semester immediately prior to enrollment and semester during enrollment in the study (approximately 5 months).
  Academic performance will be assessed using Grade Point Average (GPA). Analyses will use multilevel modeling to test for a time by condition interaction higher GPA at post treatment (and follow-up) in the equanimity compared to the strength based group.
Occurrences of Daily Acceptance | Assessed daily for seven days during week 2 and week 16 of the study.
  End-of-day perceptions of daily acceptance (used in Chin et al., under review) will be measured (Example questions" Today, I was able to accept myself as I am", "Today, I've been judging the situation that I am in or the events that are occurring as good or bad").
  Analyses will use multilevel modeling to test for a time by condition interaction showing increased acceptance and non-judgment at post-treatment in the equanimity compared to the strength based group.
Physical Activity (FitBit) | Assessed daily during week 2-17 of the study.
  Activity data for number of steps will be assessed using a FitBit device worn by participants.
  Multi-level models will test for time by treatment interactions showing increased physical activity outcomes over time in the equanimity compared to the strength based group.
Sleep (FitBit) | Assessed daily during week 2-17 of the study.
  Activity data for sleep will be assessed using a FitBit device worn by participants.
  Multi-level models will test for time by treatment interactions showing increased sleep outcomes over time in the equanimity compared to the strength based group.
Concentrations of pro-inflammatory gene expression | Change in gene expression over weeks 1 and weeks 17 of the study.
  Gene expression measures of immune system function will be collected via dried blood spot collection method.
  Multi-level models will test for time by condition effects. Analyses will focus an a priori-specified gene regulation pattern involving increased expression of inflammation-related genes and decreased expression of antiviral gene - a pattern called the conserved transcriptional response to adversity (CTRA; Cole, 2012).
Concentrations of C-Reactive Protein | Change in CRP over 4-month period.
  CRP will be assessed through dried blood spots collected at baseline and post-intervention.
  Changes in CRP will be assessed using a time by group interaction.
Concentrations of salivary cortisol | Four cortisol samples will be collected at the baseline session. One sample before and three samples after the acute stress challenge using the TSST.
  Saliva samples will be collected before and after the TSST, and assayed for salivary cortisol determination.
  Salivary cortisol will be analyzed both using area-under-the-curve (AUC) and mixed effects linear models, testing for a time by condition interaction showing that equanimity group has reduced cortisol reactivity to the TSST over time relative to the strength based group.
Perceived Stress | Change in perceived stress over 4-month period.
  Evaluated using Perceived Stress Scale (PSS). The PSS measures the degree to which situations in one's life are appraised as stressful. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress. Analyses will use multilevel modeling to test for a time by condition interaction showing decreased reported stress at post-treatment in the equanimity compared to the strength based group.
Subjective Social Status | Measured at baseline only.
  Created by health psychologist Nancy Adler and team (2000), the MacArthur Scale of Subjective Social Status is a single-item measure that assesses a person's perceived rank relative to others in their group. Respondents view a drawing of a ladder with 10 rungs, and either read that the ladder represents where people stand in society. Respondents further read : "At the top of the ladder are the people who are the best off, those who have the most money, most education, and best jobs. At the bottom are the people who are the worst off, those who have the least money, least education, worst jobs, or no job. Please place an 'X' on the rung that best represents where you think you stand on the ladder.". Rungs are translated to numbers (1-10). Choosing higher rungs of the ladder (e.g. 10) indicates perception of higher social status and choosing lower rungs of the ladder (e.g. 1) indicates lower social status.
Daily Resilience using the Brief Resilience Scale | Assessed daily for seven days during week 2 and week 16 of the study.
  End-of-day items will measure resilience over the course of the day. The Brief Resilience Scale (BRS, Smith et al. 2008) is a 6-item survey that assesses the ability to bounce back or recover from stress (e.g. "It does not take me long to recover from a stressful event."). Some items are reverse scored and then all items are summed. Higher scores reflect more resilience. Analyses will use multilevel modeling to test for a time by condition interaction showing increased resilience in daily life at post-treatment in the equanimity compared to the strength based group.
Daily Occurrence of Stress and Successful Coping Scale | Assessed daily for seven days during week 2 and week 16 of the study.
  End-of-day items will measure the perception of stress occurrence and types (e.g. "concerns about academic performance" or "family concerns") and overall perceptions of coping ability scale (e.g. Since the last survey, to what extent do you feel like your demands exceeded your ability to cope with them?") over the course of the day. Scale ranges from 0="not at all true" to 4 = "extremely true"), where higher scores indicate less successful coping (item 3 reverse scored).
  Analyses will use multilevel modeling to test for a time by condition interaction showing decreased stress (and increased coping) in daily life at post-treatment in the equanimity compared to the strength based group.
Daily State Mindfulness Scale | Assessed daily for seven days during week 2 and week 16 of the study.
  End-of-day items will measure state mindfulness over the course of the day (e.g. "I was thinking about something other than what I was currently doing" is reverse scored). The scale ranges from 0=Strongly agree to 5= Strongly disagree. Higher scores indicate higher state mindfulness.
  Analyses will use multilevel modeling to test for a time by condition interaction showing increased mindfulness in daily life at post-treatment in the equanimity compared to the strength based group.

CONTACTS AND LOCATIONS:
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kunzler AM, Helmreich I, Konig J, Chmitorz A, Wessa M, Binder H, Lieb K. Psychological interventions to foster resilience in healthcare students. Cochrane Database Syst Rev. 2020 Jul 20;7(7):CD013684. doi: 10.1002/14651858.CD013684. PMID 32691879